CLINICAL TRIAL: NCT01311505
Title: An Open Label, Single Dose, Randomized, Two-Way Cross-Over Bioequivalence Study Comparing Rifampicin In A Fixed-Dose Combination Rifampicin + Isoniazid (Myrin© 2, Pfizer Inc) Tablet With The Reference Drug (Rimactane®, Novartis Sandoz) Capsule In Healthy Filipino Male Subjects
Brief Title: Bioequivalence Study Comparing Rifampicin In A Fixed-Dose Combination (Rifampicin+Isoniazid, Myrin© 2) And The Reference Drug (Rifampicin, Rimactane®)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B3801001
Record Dates: First submitted 2011-02-15; First posted 2011-03-09 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Tuberculosis
Keywords: bioequivalence; rifampicin
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Test
  Interventions: Drug: Myrin© 2 (Rifampicin + Isoniazid)
- B (Active Comparator): Reference
  Interventions: Drug: Rimactane® (Rifampicin)

INTERVENTIONS:
Drug: Myrin© 2 (Rifampicin + Isoniazid) — Two (2) fixed-dose combination tablets each containing Rifampicin 150 mg and Isoniazid 75 mg
  Other Names: Myrin© 2 (Pfizer Inc.)
  Arms: A
Drug: Rimactane® (Rifampicin) — One (1) capsule of Rifampicin 300 mg
  Other Names: Rimactane® (Novartis Sandoz)
  Arms: B

SUMMARY:
This study is done to demonstrate bioequivalence of rifampicin component in Myrin© 2 Fixed-Dose Combination Tablet (each contains 75 mg isoniazid and 150 mg rifampicin, Pfizer Inc) with equivalent dose of the reference Rimactane® capsule (each contains 300 mg rifampicin, Novartis Sandoz) in healthy Filipino male subjects. This study also aims to determine the safety and tolerability of Myrin© 2 tablets and Rimactane® capsules in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week (1 drink = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 3 months (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* History of previous treatment for TB or is suspected of suffering from TB.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal medication, herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen / paracetamol may be used at doses of less than 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation of approximately 1 pint (500 ml) within 56 days prior to dosing.
* A history of hypersensitivity to any of the study medications or related substances, or to any of the ingredients used in the study drug formulations.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Recent history of diarrhea (2 weeks).
* Recent use of oral (2 weeks) or IV (2-3 months) antibiotics to assure normal bowel flora at study start.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Dasmariñas, Philippines

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3801001&StudyName=Bioequivalence%20Study%20Comparing%20Rifampicin%20In%20A%20Fixed-Dose%20Combination%20%28Rifampicin+Isoniazid%2C%20Myrin%A9%202%29%20And%20The%20Reference%20Drug%20%28Rifampi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 22 participants enrolled, only 21 participants were randomized since 1 participant withdrew from the study.
Groups:
- Myrin 2 First, Then Rimactane: Single oral dose of 2 fixed dose combination (FDC) tablets of Myrin 2 (each tablet contains 150 milligram (mg) rifampicin and 75 mg isoniazid) in first intervention period, and single oral dose of Rimactane capsule (300 mg rifampicin) in second intervention period. A washout period of at least 7 days was maintained between each period.
- Rimactane First, Then Myrin 2: Single oral dose of Rimactane capsule (300 mg rifampicin) in first intervention period; and single oral dose of 2 FDC tablets of Myrin 2 (each tablet contains 150 mg rifampicin and 75 mg isoniazid) in second intervention period. A washout period of at least 7 days was maintained between each period.
Period: First Intervention Period
Arm/Group | Myrin 2 First, Then Rimactane | Rimactane First, Then Myrin 2
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Washout Period (at Least 7 Days)
Arm/Group | Myrin 2 First, Then Rimactane | Rimactane First, Then Myrin 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Myrin 2 First, Then Rimactane | Rimactane First, Then Myrin 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Eligible for Analysis: Includes participants randomized to receive Myrin 2 first and Rimactane first and who had completed the study. It excludes 1 participant who did not meet the weight requirement for the study (protocol violator).
Arm/Group | Participants Eligible for Analysis
Number analyzed (Participants) | 20
Age, Customized [Number; unit: participants]
  18 to 22 years | 12
  23 to 27 years | 4
  28 to 32 years | 2
  33 to 37 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC [0-t])
Description: AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 10 hours (hrs) post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (mcg*h/mL)
Groups:
- Myrin 2: Single oral dose of 2 FDC tablets of Myrin 2 (Test) in either first intervention period or second intervention period. Each tablet contains 150 mg rifampicin and 75 mg isoniazid.
- Rimactane: Single oral dose of reference drug Rimactane capsule (300 mg rifampicin) in either first intervention period or second intervention period.
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 20 | 20
microgram*hour/milliliter (mcg*h/mL) | 38.59 (24.99) | 38.81 (21.95)
Statistical Analysis 1: Comparison: Myrin 2 vs Rimactane; 20 participants (10 per sequence) provided at least 98% power that 90% confidence interval (CI) for ratio of test to reference for AUC(0-t) of rifampicin lie within acceptance region of 80%-125%. Intra-participant coefficient of variation (CV) estimate of approximately 13.48% for AUC(0-t) was used for this power calculation. Natural log transformed AUC(0-t) was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; Ratio of adjusted geometric means = 98.90, 90% CI 2-sided [92.98 to 105.20]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 10 hrs post-dose
Population: PK parameter analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Rimactane: Single oral dose of reference drug Rimactane capsule (300 mg capsule) in either first intervention period or second intervention period.
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 20 | 20
mcg/mL | 7.89 (24.89) | 8.02 (22.35)
Statistical Analysis 1: Comparison: Myrin 2 vs Rimactane; 20 participants (10 per sequence) provided at least 94% power that 90% CI for ratio of test to reference for Cmax of rifampicin lie within acceptance region of 80%-125%. Intra-participant CV estimate of approximately 16.43% for Cmax was used for this power calculation. Natural log transformed Cmax was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as random effect; Test type: Superiority or Other; Ratio of adjusted geometric means = 98.24, 90% CI 2-sided [87.77 to 109.97]

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 10 hrs post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hrs
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 20 | 20
hrs | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]

4. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0-∞])
Description: AUC (0-∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 10 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 20 | 20
mcg*hr/mL | 47.72 (30.54) | 47.15 (25.32)
Statistical Analysis 1: Comparison: Myrin 2 vs Rimactane; Natural log transformed AUC(0-∞) of rifampicin was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Ratio of adjusted geometric means = 100.25, 90% CI 2-sided [94.44 to 106.41]

5. Secondary Outcome: Plasma Decay Half-life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 10 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 20 | 20
hrs | 4.0750 (1.0777) | 3.8635 (0.8347)

6. Secondary Outcome: Extrapolated Area Under the Curve (AUC Percent [%] Extrapolated)
Description: AUC%extrapolated is the extrapolated area under the plasma concentration time profile following the last measured concentration. It is calculated as (AUC [0-∞] minus AUC[0-10])*100/ AUC (0-∞), where AUC (0-∞) = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-∞) and AUC(0-10) = area under the plasma concentration time-curve from zero (pre-dose) to the last quantifiable concentration.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 and 10 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent AUC
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 20 | 20
Percent AUC | 18.84 (38.47) | 17.53 (30.23)

7. Other Pre Specified Outcome: Number of Participants With Abnormal Safety Laboratory Test Values
Description: Participants were evaluated for following safety laboratory tests: Hematology, chemistry, urinalysis.
Time Frame: Screening and Follow-up (1 week post-baseline)
Population: Safety population included participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Myrin 2: Single oral dose of 2 FDC tablets of Myrin 2 (Test) in either first intervention period or second intervention period. Each tablet contains 150 rifampicin and 75 mg isoniazid.
- Rimactane: Single oral dose of reference drug Rimactane 300 mg capsule in either first intervention period or second intervention period.
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 20 | 21
participants
  Screening | 0 | 0
  Follow-up | 0 | 0

8. Other Pre Specified Outcome: Clinically Significant Change From Baseline Supine Blood Pressure (BP)
Description: Mean change: vital sign value at observation (Day 1 and follow-up) minus vital sign value at baseline.
Time Frame: Baseline (Day 0), Day 1 (Hour 10), and follow-up (1 week post-baseline)
Population: Data was not summarized since supine systolic and diastolic BP remained within normal limits throughout the study and there were no significant deviations from baseline.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Clinically Significant Change From Baseline Pulse Rate
Description: Mean change: vital sign value at observation (Day 1 and follow-up) minus vital sign value at baseline.
Time Frame: Baseline (Day 0), Day 1 (Hour 10), and follow-up (1 week post-baseline)
Population: Data was not summarized since pulse rate remained within normal limits throughout the study and there were no significant deviations from baseline.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Clinically Significant Change From Baseline Oral Temperature
Description: Mean change: vital sign value at observation (Day 1 and follow-up) minus vital sign value at baseline.
Time Frame: Baseline (Day 0), Day 1 (Hour 10), and follow-up (1 week post-baseline)
Population: Data was not summarized since oral temperature remained within normal limits throughout the study and there were no significant deviations from baseline.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Clinically Significant Change From Baseline Respiratory Rate
Description: Mean change: vital sign value at observation (Day 1 and follow-up) minus vital sign value at baseline.
Time Frame: Baseline (Day 0), Day 1 (Hour 10), and follow-up (1 week post-baseline)
Population: Data was not summarized since respiratory rate remained within normal limits throughout the study and there were no significant deviations from baseline.
Measure: Mean (Standard Deviation); unit: respirations/minute
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: Any untoward medical occurrence in a participant who received study treatment was considered an AE without regard to possibility of causal relationship.
Time Frame: Baseline (Day 0), Day 1 and Follow-up (1 week post-baseline)
Population: Safety population included participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Myrin 2 | Rimactane
Number analyzed (Participants) | 20 | 21
participants
  Day 0 | 0 | 0
  Day 1 | 0 | 0
  Follow-up | 0 | 0

ADVERSE EVENTS:
Arm/Group | Myrin 2 | Rimactane
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes